CLINICAL TRIAL: NCT03265275
Title: Why Still in Hospital After Hip Fracture Surgery?
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Asbjorn Aroen, Professor, University Hospital, Akershus
Other Study IDs: 2017/CP
Record Dates: First submitted 2017-08-23; First posted 2017-08-29 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Hip Fractures
Keywords: Fast track
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fast track patient pathway — Prehospital services establish a working diagnosis of hip fracture and initiate first line treatment. In the emergency department a specially trained nurse triages the patient. Patients without signs of other acute disease or trauma and who have not previously been operated in the same hip are directly transported to the x-ray suite. The x-rays are reviewed by the radiographer and in case of an obvious fracture of the hip the patient is transported directly to the orthopedic ward where the patient is received by a nurse and seen by an orthopedic surgeon. The pathway includes standard procedures for blood sampling, pain relief, including a fascia iliaca compartment block, intravenous fluids, transfusion triggers, management of anticoagulants and premedication. The pathway puts focus on prevention of pressure sores, a short preoperative fasting period and early mobilization. Screening tools are used to assess for delirium, nutritional status and fall risk.

SUMMARY:
At our institution, hip fracture patients are admitted and treated according to a fast track patient pathway. The aim of this study is to identify areas of this patient pathway that can be improved. To achieve this, the study will investigate the underlying reasons for the continued need for hospitalization on the consecutive days after hip fracture surgery.

DETAILED DESCRIPTION:
The study will be conducted at the orthopedic department, Akershus University Hospital, as a prospective observational study and will include approximately 200 consecutive hip fracture patients. The patients will be evaluated once daily for the fulfillment of predefined discharge criteria. If the discharge criteria are not met or if the criteria are met but the patient is not discharged in spite of this the underlying reason(s) are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Operated at the orthopedic department, Akershus University Hospital, for a hip fracture

Exclusion Criteria:

* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, who have been operated for a hip fracture at the orthopedic department, Akershus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Factors necessitating hospitalization after hip fracture surgery | Recorded using a check-list once daily from first day after hip fracture surgery until discharge from the orthopedic department, typically between 1 to 14 days after hip fracture surgery
  Recorded as: acute anemia, delirium, medical complications, pain, dizziness, nausea/vomiting, logistical reasons, unwillingness to be discharged, other (specified as free text)

SECONDARY OUTCOMES:
Percentage of patients discharged to their preoperative level of care | At hospital discharge, typically between 1 to 14 days after hip fracture surgery
Length of hospital stay | At hospital discharge, typically between 1 to 14 days after hip fracture surgery
  Length of hospital stay in days, stratified after type of operation

CONTACTS AND LOCATIONS:
Overall Officials: Asbjorn Aaroen, Professor, Study Director — University Hospital, Akershus
Locations (1):
- Akershus University hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No